CLINICAL TRIAL: NCT07344961
Title: Determinates of Atrial Tracking and Prevalence of Atrial Fibrillation in the Micra AV2 (DANCE AFIB)
Acronym: DANCE AFIB
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 25-0696; 0696 (Other: Northwell)
Record Dates: First submitted 2025-12-10; First posted 2026-01-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Micra AV2- Observational — All eligible patients that have a history of paroxysmal atrial fibrillation and an indication to undergo Micra AV2 device placement as per standard of care (SOC) across the participating sites within the Northwell Health System can be included in this analysis. Micra AV2 placement indications will be at the discretion of the treating electrophysiologist, but are expected to be predominantly atrioventricular block.

SUMMARY:
This is a prospective, descriptive study. Safety endpoints will not be assessed. All eligible patients that have a history of paroxysmal atrial fibrillation and an indication to undergo Micra AV2 device placement as per standard of care (SOC) across the participating sites within the Northwell Health System can be included in this analysis. Micra AV2 placement indications will be at the discretion of the treating electrophysiologist, but are expected to be predominantly atrioventricular block. Periodic device interrogations will be reviewed for the presence of effective atrial tracking during sinus rhythm . The presence of paroxysmal atrial fibrillation and the degree to which atrial activity and A4 amplitude trend changes will be assessed using a designated Medtronic Research Holter monitor that detects Micra AV2 signals at any point in the study during a episodes of sinus rhythm and atrial fibrillation. Patients who have atrial fibrillation during index hospitalization will undergo placement of the Medtronic Holter monitor as part of the standard of care index hospitalization. Eligible outpatients will undergo placement of the Medtronic Research Holter Monitor in the office.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legally authorized representative (LAR) provides authorization and/or consent per institution and geographical requirements
* Participant has been implanted with the Micra AV2 device or is intended to receive or be treated with an eligible Micra AV2 device as per standard of care.
* Participants with a history of paroxysmal atrial fibrillation undergoing Micra AV2 implantation, as per standard of care.
* Age 18-85 years old with the ability to consent for the procedure
* Participant is consented within the enrollment window of the therapy received, as applicable
* English Speaking

Exclusion Criteria:

* Participant who is, or is expected to be, inaccessible for follow-up
* Participation is excluded by local law
* Participant is currently enrolled or plans to enroll in concurrent drug/device study that may confound the study results
* Participant with persistent/chronic atrial fibrillation
* Prisoner or cognitively impaired due to the study procedures involving independent wearing of the holter monitor for research purposes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: AFIB patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the prevalence of atrial fibrillation in the Micra AV2 patients | Through study completion, an average of 6 months
To evaluate A4 amplitude trend changes during sinus rhythm and atrial fibrillation | Through study completion, an average of 6 months
  To evaluate the presence of paroxysmal atrial fibrillation and the degree to which atrial activity and A4 amplitude trend changes will be assessed using a designated Medtronic Research Holter monitor that detects Micra AV2 signals at any point in the study during episodes of sinus rhythm and atrial fibrillation.
To determine the ability of the Micra AV2 device to detect the presence and burden of atrial fibrillation | Through study completion, an average of 6 months
  Micra AV2 placement indications will be at the discretion of the treating electrophysiologist, but are expected to be predominantly atrioventricular block. Periodic device interrogations will be reviewed for the presence of effective atrial tracking during sinus rhythm.

CONTACTS AND LOCATIONS:
Overall Officials: Haisam Ismail, MD, Principal Investigator — Northwell Health
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No